CLINICAL TRIAL: NCT05622968
Title: Outpatient Cervical Ripening With Foley Catheter for Induction of Labour in Low Risk Women: a Quasi-experimental Study (OFC Study)
Brief Title: Outpatient Induction of Labour Using Intracervical Foley Catheter
Acronym: OFC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: Hospital Kemaman (Other)
Responsible Party: Principal Investigator, Zahar Azuar Zakaria, Principal Investigator, Head of Obstetric & Gynecology Department, Senior Consultant, Hospital Kemaman
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMRR ID-22-00349-EQQ
Record Dates: First submitted 2022-11-14; First posted 2022-11-21 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Pregnancy Related; Induction of Labor Affected Fetus / Newborn
Keywords: outpatient induction; Foley catheter
MeSH Terms: interventions — Urinary Catheters; Dinoprostone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Active Comparator): Women who are planned for elective delivery for obstetric indication(s) and undergo outpatient induction of labour using Foley catheter
  Interventions: Device: Foley catheter; Drug: Intravaginal prostaglandin E2
- Control (Placebo Comparator): Women who are planned for elective delivery for obstetric indication(s) and undergo inpatient induction of labour using intravaginal prostaglandin
  Interventions: Drug: Intravaginal prostaglandin E2

INTERVENTIONS:
Device: Foley catheter — Insertion of 18G Foley catheter into the cervical canal and inflating the balloon to 60 mls using sterile water
  Other Names: urinary catheter
  Arms: Intervention
Drug: Intravaginal prostaglandin E2 — Insertion of intravaginal Dinoprostone
  Other Names: Dinoprostone

SUMMARY:
Prospective quasi-experimental study between a study population who will receive outpatient induction of labour using intracervical Foley catheter, followed by the inpatient induction using intravaginal prostaglandin and a control group of women with similar characteristics undergoing inpatient labour induction with intravaginal prostaglandin (standard management)

DETAILED DESCRIPTION:
The study will be conducted among pregnant women in 2 to 5th pregnancy who have no significant risk factors and planned for induction of labour. The eliiable women will be recruited from 4 health clinics within the district (of Kemaman, Malaysia) and located within 20 km from the hospital.

Willing participants will be seen in the hospital at the planned induction date and reassessed. Should they be suitable for induction of labour using Foley catheter on outpatient basis, a 18G Foley catheter will be inserted into the cervical canal and the balloon inflated with sterile water (60 mls). The fetal well being will be assessed and the women allowed to go home with instruction related to the induction and the study.

Those who do not enter the active phase of labour will be admitted to the ward 24 hours later and will undergo inpatient induction of labour using intravaginal prostaglandin (Dinoprostone) according to the local protocol.

These women will be compared with a control group comprising of women with similar characteristics and undergo inpatient induction of labour with intravaginal Dinoprostone.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 year old
* Singleton pregnancy
* Cephalic presentation
* Multiparous women in their 2nd to 5th pregnancy (Para 1 to 4)
* Gestational age between 37+0 and 41+0 weeks.
* No previous uterine surgery (lower segment caesarean section, upper segment caesarean section, myomectomy
* Resides within 30 minutes drive from Hospital Kemaman
* Has access to a telephone
* Has reliable transportation (i.e. able to get to the hospital immediately without the need of ambulance)
* Acceptance of participation by the signing of a written consent.

Exclusion Criteria:

* Pregnancy with non-cephalic presentation
* Prior cesarean delivery
* Gestational hypertension or preeclampsia on 2 or more medications
* Diabetes in pregnancy on high dose medication(s); insulin of more than 60 units per day or combination of insulin and oral hypoglycemic agent
* Low lying placenta or placenta praevia
* Rupture of amniotic membrane
* Primiparae and grandmultiparae (para 5 or more)
* Multiple pregnancy
* Fetal death
* Fetal anomalies: defined as the presence of a major fetal anomaly of any organ system
* Fetal growth restriction: defined as an ultrasound derived estimated fetal weight less than the 10th percentile for gestational age
* Suspected macrosomia: defined as an ultrasound derived estimated fetal weight of more than 90th centile for gestational age
* Oligohydramnios: ultrasound measured amniotic fluid index (AFI) less than the 10th percentile for gestational age
* Polyhydramnios: defined as an AFI of 24 cm or greater or a single deepest vertical pocket of 8 cm or greater
* Latex allergy
* Contraindication to induction of labor
* Evidence of active phase of labor

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — All low risk pregnant women with obstetric indication for induction of labour at term
Enrollment: 88 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Induction of labour-delivery interval | Induction of labour (intravaginal prostaglandin) to delivery
  The mean interval between the start of inpatient cervical ripening and delivery (from the start of cervical ripening with Dinoprostone to the delivery of the baby)

SECONDARY OUTCOMES:
Success rate of induction of labour within 12 hours | From the start of inpatient cervical ripening and delivery
  The percentage of vaginal delivery within 12 hours of inpatient cervical ripening
Success rate of induction of labour within 24 hours | From the start of inpatient cervical ripening and delivery
  The percentage of vaginal delivery within 24 hours of inpatient cervical ripening
Delivery outcome | Induction to delivery
  Percentage of caesarean section and instrumental delivery
Adverse event | Induction to delivery
  Incidence of uterine tachysystole and hyperstimulation
Labour augmentation | Induction to delivery
  Duration and maximum oxytocin dose used for labour augmentation
Maximum pain recorded | Induction to delivery
  Maximum recorded contraction pain during cervical ripening (using Visual Analogue Scale of 10)
Incidence of chorioamnionitis | Induction to 24 hours after delivery
  maternal temperature is greater than or equal to 39.0°C or when the maternal temperature is 38.0-38.9°C and one additional clinical risk factor is present
Analgesia requirement | Induction to delivery
  Prevalence of analgesia required during induction of labour
Postpartum hemorrhage | Delivery to 24 hours after delivery
  Primary postpartum haemorrhage (blood loss of more than 500mls within 24 hours of delivery)
Neonatal Apgar score | Delivery to 10 minutes after birth
  Incidence of low Apgar score (less than 7) at 5 minutes after delivery
Neonatal intubation | Delivery to 30 minutes after birth
  Incidence of neonates requiring intubation
Neonatal seizure | Delivery to 24 hours after birth
  Incidence of neonate with seizure
Neonatal complication | Delivery to 24 hours after birth
  Admission to the Neonatal Intensive Care Unit

CONTACTS AND LOCATIONS:
Overall Officials: Zahar Zakaria, MD, Principal Investigator — Hospital Kemaman
Locations (1):
- Hospital Kemaman, Kampong Kemaman, Terengganu, Malaysia

IPD SHARING:
Plan to Share IPD: No
No plan to share for now

REFERENCES:
- [Background] Sharp AN, Stock SJ, Alfirevic Z. Outpatient induction of labour in the UK: a survey of practice. Eur J Obstet Gynecol Reprod Biol. 2016 Sep;204:21-3. doi: 10.1016/j.ejogrb.2016.06.023. Epub 2016 Jul 30. PMID 27513897
- [Result] Royal College of Obstetricians and Gynaecologists. Evidence-based Clinical Guideline No. 9. Induction of labour
- [Result] ACOG Practice Bulletin No. 107: Induction of labor. Obstet Gynecol. 2009 Aug;114(2 Pt 1):386-397. doi: 10.1097/AOG.0b013e3181b48ef5. No abstract available. PMID 19623003
- [Result] Leduc D, Biringer A, Lee L, Dy J; CLINICAL PRACTICE OBSTETRICS COMMITTEE; SPECIAL CONTRIBUTORS. Induction of labour. J Obstet Gynaecol Can. 2013 Sep;35(9):840-857. doi: 10.1016/S1701-2163(15)30842-2. English, French. PMID 24099451
- [Result] Dowswell T, Kelly AJ, Livio S, Norman JE, Alfirevic Z. Different methods for the induction of labour in outpatient settings. Cochrane Database Syst Rev. 2010 Aug 4;(8):CD007701. doi: 10.1002/14651858.CD007701.pub2. PMID 20687092
- [Result] Vogel JP, Osoti AO, Kelly AJ, Livio S, Norman JE, Alfirevic Z. Pharmacological and mechanical interventions for labour induction in outpatient settings. Cochrane Database Syst Rev. 2017 Sep 13;9(9):CD007701. doi: 10.1002/14651858.CD007701.pub3. PMID 28901007
- [Result] Dong S, Khan M, Hashimi F, Chamy C, D'Souza R. Inpatient versus outpatient induction of labour: a systematic review and meta-analysis. BMC Pregnancy Childbirth. 2020 Jun 30;20(1):382. doi: 10.1186/s12884-020-03060-1. PMID 32605542
- [Result] Croll DMR, Hoge PC, Verhoeven CJM, de Boer MA, Bloemenkamp KWM, de Heus R. Changes in local protocols on inpatient cervical priming and introduction of outpatient priming: A nationwide survey in the Netherlands. Eur J Obstet Gynecol Reprod Biol. 2021 Aug;263:148-152. doi: 10.1016/j.ejogrb.2021.06.004. Epub 2021 Jun 10. PMID 34214801
- [Result] Amorosa JM, Stone JL. Outpatient cervical ripening. Semin Perinatol. 2015 Oct;39(6):488-94. doi: 10.1053/j.semperi.2015.07.014. Epub 2015 Sep 11. PMID 26365009
- [Result] Kruit H, Heikinheimo O, Ulander VM, Aitokallio-Tallberg A, Nupponen I, Paavonen J, Rahkonen L. Foley catheter induction of labor as an outpatient procedure. J Perinatol. 2016 Aug;36(8):618-22. doi: 10.1038/jp.2016.62. Epub 2016 Apr 14. PMID 27078202
- [Result] Sciscione AC, Muench M, Pollock M, Jenkins TM, Tildon-Burton J, Colmorgen GH. Transcervical Foley catheter for preinduction cervical ripening in an outpatient versus inpatient setting. Obstet Gynecol. 2001 Nov;98(5 Pt 1):751-6. doi: 10.1016/s0029-7844(01)01579-4. PMID 11704164
- [Result] Diederen M, Gommers J, Wilkinson C, Turnbull D, Mol B. Safety of the balloon catheter for cervical ripening in outpatient care: complications during the period from insertion to expulsion of a balloon catheter in the process of labour induction: a systematic review. BJOG. 2018 Aug;125(9):1086-1095. doi: 10.1111/1471-0528.15047. Epub 2018 Jan 10. PMID 29211328
- [Result] Stephenson E, Borakati A, Simpson I, Eedarapalli P. Foley catheter for induction of labour: a UK observational study. J Obstet Gynaecol. 2020 Nov;40(8):1064-1068. doi: 10.1080/01443615.2019.1676213. Epub 2019 Dec 3. PMID 31793372
- [Result] Turnbull D, Adelson P, Oster C, Bryce R, Fereday J, Wilkinson C. Psychosocial outcomes of a randomized controlled trial of outpatient cervical priming for induction of labor. Birth. 2013 Jun;40(2):75-80. doi: 10.1111/birt.12035. Epub 2013 Mar 25. PMID 24635460